CLINICAL TRIAL: NCT02804594
Title: A Phase 2 Randomized, Placebo- Controlled, Parallel Group, Double Blinded Single Center Study on Effect of N-acetyl Cysteine Compared to Placebo on Fatigue in Patients With Progressive Multiple Sclerosis
Brief Title: A Study of Oxidative Pathways in MS Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAC Pilot
Record Dates: First submitted 2016-06-03; First posted 2016-06-17 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Progressive Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Fatigue | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetyl cysteine (Active Comparator): 1250 mg of N-acetyl cysteine three times daily
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): placebo three times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — 1250 mg of N- acetyl cysteine taken three times daily
  Other Names: NAC
  Arms: N-acetyl cysteine
Drug: Placebo — placebo taken three times daily
  Arms: Placebo

SUMMARY:
This is a 4-week randomized, placebo-controlled, parallel group, double-blind, single center trial on effect of N-acetyl cysteine versus placebo on fatigue in patients with progressive MS defined by McDonald criteria. Subjects who enter the treatment phase of study, will be randomly assigned to either N-acetyl cysteine (1250 mg three times a day) or placebo (three times a day) for 4 weeks. There will be 3 in-person study visits (screening, baseline, and week 4) and 2 visits over the phone (week 2, and week 6 which is 2 weeks after completing last study drug dose). Visits will all occur in the morning to maximize consistency of assessments and evaluate main outcomes within 2 hours of morning dose of study medication. Fatigue questionnaires, and research samples will be obtained before neurological examination, or magnetic resonance imaging. Research blood draws will be obtained just after fatigue questionnaire completion. Brain spectroscopy will be obtained less than 2 hours after morning dose of study drug to maximize detection of the biological effect of study medication.

DETAILED DESCRIPTION:
1Background 1.1 Multiple Sclerosis Multiple sclerosis is the most common cause of non-traumatic disability in young adults in the US. It is an inflammatory, demyelinating and neurodegenerative disease of the central nervous system. Patients with MS often experience various types of disabling symptoms such as chronic fatigue or pain. Most patients with an initial relapsing-remitting course develop at some point insidious disability worsening, i.e. secondary progressive MS. In contrast, about 15% of multiple sclerosis patients experience an insidiously progressive course from onset. Primary and secondary progressive multiple sclerosis is thought to have similar physiopathology. As such, strategies for managing symptoms of relapsing patients may not necessarily apply to those with progressive disease; however, most symptomatic treatment trials have been done in relapsing-remitting or mixed populations of patients, neglecting a large fraction of patients with progressive forms of the disease. Investigator is planning to address an important clinical and pathophysiologic issue in this proposed study.

1.2 Fatigue in multiple sclerosis Fatigue as defined by a subjective lack of physical or mental energy perceived by the individual with usual activities is the most common and disabling symptom of multiple sclerosis. Fatigue severity is not correlated with depression or neurological disability. It can impact substantially physical and cognitive activities and thus, negatively affect the quality of life of many patients. There are no medications specifically approved for fatigue in multiple sclerosis. Many chronic inflammatory disorders are associated with fatigue and peripheral inflammation is postulated to be an important contributor to fatigue pathogenesis. A spectroscopy study has reported decreased N-acetylaspartate/creatine ratio in several brain regions, thus all pointing at axonal loss as a possible contributing factor . In a cross-sectional relapsing-remitting MS study, fatigued patients had more severe atrophy of the striatum, thalamus and frontal and parietal gyri as compared to non-fatigued patients.

As a direct consequence of the unknown pathophysiology, very little pharmacologic intervention is available for fatigue in multiple sclerosis. Glutamate, a critical neurotransmitter implicated in excitotoxicity and neurodegeneration, may also play a role in fatigue genesis. Two studies of a glutamate receptor antagonist (memantine) have reported worsening of fatigue in multiple sclerosis patients. In addition, Investigator have found that compared to placebo, riluzole (a medication with some anti-glutamate activity) worsened fatigue in patients with very early multiple sclerosis. This is in sharp contrast with the pathological evidence suggesting that excessive glutamate transmission may be a final effector in neuronal and axonal degeneration in multiple sclerosis animal models. Oxidative stress due to disequilibrium between oxidants and antioxidants in the central nervous system may also be a major contributor to neurodegeneration . It is unknown if oxidative stress plays a role in the pathogenesis of fatigue in multiple sclerosis.

1.3 Fatigue rating scales Most of the fatigue scales used in multiple sclerosis studies were primarily developed and validated for use in other medical conditions. The two widely used self-completed scales in multiple sclerosis research are the Fatigue Severity Scale, and the Modified Fatigue Impact Scale.

1.3a. Fatigue Severity Scale: This scale was originally designed to identify the common features of fatigue in multiple sclerosis, and lupus patients. It assesses the impact of fatigue on several outcomes, with an emphasis on physical fatigue. It is composed of 9 questions with responses provided on a 7-point Likert scale. Scale score is the mean of the item scores and higher scores indicate more severe fatigue.

1.3b.Modified Fatigue Impact Scale: This scale has been proposed by the Multiple Sclerosis Council for Clinical Practice Guidelines as the instrument of choice for assessing fatigue in multiple sclerosis. It is derived from the 40-item Fatigue Impact Scale. It has 21 items and assesses more dimensions of fatigue than the Fatigue Severity Scale: physical (9 items), cognitive (10 items) and psychosocial (2 items). The scale score is the sum of the 21 items and higher score indicates more severe fatigue. The scale has shown good reproducibility, ease of use and good correlation with fatigue severity scale scores. A cut-off value of 38 distinguishes fatigued from non-fatigued multiple sclerosis patients.

2.Rationale 2.1 Effect of N-acetyl cysteine in MS fatigue N-acetyl cysteine is an orally bioavailable precursor of the amino acid cysteine and is used to treat acetaminophen-induced hepatotoxicity. The medication half-life in adults is about 5.6 hours. As such it has been given twice or three times a day in various trials that have documented a biological effect. It protects the liver by restoring hepatic concentrations of cysteine and glutathione (GSH- a major intracellular antioxidant). Besides antioxidant properties, N-acetyl cysteine, by increasing the intracellular concentration of cysteine and activating the glutamate-cysteine antiporter eventually decreases glutamatergic transmission. Hypothetically, by decreasing excitotoxicity, it may protect neurons in different models of neuronal damage and neurodegeneration. Excellent safety profile and potential neuroprotective properties make N-acetyl cysteine an attractive target for examining its anti-fatigue properties in patients with progressive multiple sclerosis. Orally administered N-acetyl cysteine produces biologically relevant cerebrospinal fluid concentrations of N-acetyl cysteine at doses that are well tolerated. One study showed an effect of a single injection of N-acetyl cysteine on blood glutathione redox ratios followed by changes in glutathione concentration in the brain using 7T magnetic resonance spectroscopy in 3 patients with Parkinson's disease and 3 controls.

Clinical trials of oral N-acetyl cysteine for a wide variety of clinical conditions have used a range of different daily doses (from 600 mg to 6000 mg per day). The study investigator chose the daily dose of 3750 mg (1250 mg administered three times a day), based on its good tolerability, treatment compliance and minimum adverse effects reported in a recent clinical trial.

2.2 Reason for using a placebo group

There are no FDA-approved treatments for fatigue in multiple sclerosis. There are also no standard of care as various trials have reported inconsistent findings about the effect of amantadine in multiple sclerosis fatigue. Pursuant to the Helsinki Declaration, when standard treatment of a disease exists, placebo should generally not be used in clinical trials. However, Declaration of Helsinki supports the stance that placebo can be acceptable in the setting where no proven standard therapy exists:

The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:

* The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
* Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm.

2.3 Gap in fatigue management Symptomatic treatment trials for fatigue have been small, underpowered and with methodological flaws. As such, drawing firm conclusions and making therapeutic recommendations has been difficult. Thus, fatigue in multiple sclerosis remains very difficult to manage despite its substantial impact on patients' life. An issue when studying fatigue in patients with relapsing-remitting multiple sclerosis has been the possibility of increased fatigue during disease relapses and with specific disease-modifying therapies such as interferon. There has been no study focusing on the effects of drug therapy in fatigue in patients with progressive disease. Furthermore, study investigator's knowledge regarding the underlying pathophysiology of fatigue in multiple sclerosis is scarce and future studies of intervention on fatigue should include biomarkers to further elucidate the potential mechanisms of observed effects.

The study investigator hypothesize that fatigue in progressive multiple sclerosis patients is associated with increased glutamate and decreased glutathione concentration on brain spectroscopy at baseline. The study investigator also hypothesize that fatigue is associated with changes of various oxidative pathway metabolites in peripheral blood.

4. Study Design 4.1 Overview of study design: This is a 4-week randomized, placebo-controlled, parallel group, double-blind, single center trial on effect of N-acetyl cysteine versus placebo on fatigue in patients with progressive multiple sclerosis defined by McDonald criteria. Subjects, who enter the treatment phase of study, will be randomly assigned to either N-acetyl cysteine (1250mg 3 times a day or placebo ( three times a day)for 4 weeks.There will be 3 in-person study visits (screening, baseline, and week 4 and 2 visits over the phone (week 2, and week 6 which is 2 weeks after completing last study drug dose). Visits will all occur in the morning to maximize consistency of assessments and evaluate main outcomes within 2hours of morning dose of study medication. Questionnaires, and research samples will be obtained before neurological exam or magnetic resonance imaging. Research blood draws will be obtained just after questionnaire completion. Brain spectroscopy will be obtained less than 2hours after morning dose of study drug to maximize detection of the biological effect of study medication.

4.2 Enrollment sites Enrollment will start in August, 2016. Enrollment period will last 6 months. Patients will be enrolled in the trial at University of California San Francisco.

4.3 Study visits 4.3a Screening period: Total duration of screening period is 4 weeks. An additional 5 patients with progressive multiple sclerosis who volunteered for participation in the clinical trial, but had a screening modified fatigue impact scale score of <38 or were recruited from site's clinic (who reported no fatigue and their fatigue scale score was <38), will undergo brain imaging on 7Tesla magnetic resonance imaging machine, and research blood draws.

4.3b Treatment period: Total duration of the blinded treatment period is 4 weeks. After the screening visit, the inclusion/ exclusion criteria details of eligible patients will be reviewed by study investigator. The eligible study participants will be randomized in approximately a 2:1 ratio to one of the two arms of either N-acetyl cysteine or placebo. The treatment group assignment will be blinded for the duration of the study. A week-2 phone visit will be completed to determine the tolerance of study drug.

4.3c Follow up phone visit: Two weeks after taking the last dose of study medication, fatigue scale questionnaires are completed over phone by the study coordinator to collect the safety and efficacy measures of the study. Additional phone visit needs to be completed 2 weeks from randomization to assess the safety, tolerability, and compliance of study medication.

4.5 Study visit window: The screening period can be up to 4 weeks. The baseline visits needs to be completed within 28 days of screening visit. Week 2 phone visit in +/- 5 days of Day 14, and week 4visit in Day 28+/-7 days of baseline. Follow-up phone call is completed +/- 5 days of week 6 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 75 years included.
2. Ability to sign the informed consent before participation.
3. Females of childbearing age must have a negative pregnancy test at screening and use an effective method of contraception during the study participation period.
4. Diagnosis of primary or secondary progressive multiple sclerosis (according to the 2010 McDonald criteria).
5. Time since first reported MS symptoms more than one year.
6. EDSS score at the time of screening 2.0-6.5.
7. Fatigue reportedly present and screening MFIS more than 38 for patients who will be enrolled in the randomized placebo controlled part of the study. MFIS score of less than 38 is required for patients who are controls on the study.

Exclusion Criteria:

1. History of MS relapses in the previous 3 months.
2. Neurodegenerative progressive neurological disorders other than progressive MS.
3. Breastfeeding
4. History of bleeding disorders
5. Abnormal results of liver function test at screening (AST or ALT more than twice the upper limit of normal).
6. Receiving or about to start interferon beta or immunosuppressive medications (e.g. cyclophosphamide, mitoxantrone, methotrexate, mycophenolate mofetil) as these medication can be associated with fatigue.
7. Starting or changing the dose of other MS disease-modifying medications (including monoclonal antibodies such as rituximab, ocrelizumab, alemtuzumab, daclizumab) within 3 months of baseline visit.
8. No ongoing steroid treatment and no steroid treatment in the prior month.
9. Inability to undergo MRI scans (e.g. weight>350 pounds, severe claustrophobia, metal in the body).
10. Medical terminal conditions.
11. Currently treated for active malignancy or metastatic malignancy that has been treated in the past 1 year or undergoing extra screening for recurrence
12. Planned surgery within the following 12 weeks
13. Planning to move with the following next 12 weeks
14. Participating in another clinical trial with an experimental medication.
15. Alcohol or substance abuse, or any other condition that in the investigator's opinion would make the patient unsuitable for this study.
16. A history of allergic or anaphylactic reaction to NAC, or any component of the preparation.
17. Clinically unstable medical or psychiatric disorders that require acute treatment.
18. Active gastrointestinal ulcers.
19. Subjects taking concomitant medications or supplements known for their glutamatergic effects (e.g., dextromethorphan, D-cycloserine, memantine, lamotrigine, riluzole), antioxidant properties (DMG, TMG, other alternative treatments), or medications with an effect on sleepiness and possibly fatigue such as Provigil, Nuvigil and amantadine within 2 weeks of the baseline visit with the exception of short-term use of dextromethorphan as needed as a cough suppressant. Regular multivitamins will be allowed.
20. Patients taking anticoagulants
21. Patients with history of obvious secondary causes of fatigue, such as chronic insomnia, sleep apnea, narcolepsy, restless leg syndrome and significant bladder dysfunction disrupting sleep.
22. Screening Epworth Sleepiness Scale score greater than 15.
23. Starting or changing the dose of benzodiazepine, antidepressant, antipsychotics, anti-histamines, or stimulants within a month from the screening visit.
24. A score of 15 or greater on the Hospital Anxiety and Depression Scale (HADS) depression subscale.
25. Patients currently treated for asthma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Waubant, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krysko KM, Bischof A, Nourbakhsh B, Henry RG, Revirajan N, Manguinao M, Nguyen K, Akula A, Li Y, Waubant E. A pilot study of oxidative pathways in MS fatigue: randomized trial of N-acetyl cysteine. Ann Clin Transl Neurol. 2021 Apr;8(4):811-824. doi: 10.1002/acn3.51325. Epub 2021 Mar 6. PMID 33675156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our study participants are recruited from the MS Clinic.
Pre-assignment Details: Study participants who met the eligibility criteria to enroll in the study are randomized into study medication group or placebo group. Study participants who did not meet the criteria to enter the study treatment period of the study were observed as controls.
Period: Overall Study
Arm/Group | N-acetyl Cysteine | Placebo
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetyl Cysteine | Placebo | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 11
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (9.2) | 65.7 (6.8) | 56.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 5 | 15
Modified Fatigue Impact Scale (MFIS) score at baseline [Median (Inter-Quartile Range); unit: Scores on a scale] — The MFIS is a self-report measure to rate fatigue in Multiple Sclerosis. The total score, ranging from 0 to 84 is the sum of three subscales (physical, cognitive, and psychosocial functioning). Higher numbers indicate greater fatigue. Modified fatigue Impact scale of more than 38 is one of the inclusion criteria for the study.
  Scores on a scale | 48.5 [46 to 56] | 50 [45 to 52] | 50 [45 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported Since Baseline Visit That Are Related to N-acetyl Cysteine.
Description: Number of adverse events reported since baseline visit that are related to N-acetyl cysteine will be compared to the number of adverse events reported by participants in the placebo group.
Time Frame: 4 weeks
Population: Study participants enrolled in the treatment period are included in the analysis.
Measure: Number; unit: adverse events
Arm/Group | N-acetyl Cysteine | Placebo
Number analyzed (Participants) | 10 | 5
adverse events | 12 | 6

2. Secondary Outcome: Change in Fatigue Score on Questionnaires From Baseline
Description: Change in fatigue score on questionnaires from baseline visit to week-4 is calculated for the Modified Fatigue Impact Scale (MFIS) questionnaire. The MFIS is a self-report measure to rate fatigue in Multiple Sclerosis. The total score, ranging from 0 to 84 is the sum of three subscales (physical, cognitive, and psychosocial functioning). Higher numbers indicate greater fatigue. Modified fatigue Impact scale of more than 38 is one of the inclusion criteria for the study. Study participants who scored higher value on the questionnaire at week-4 are considered to have worsened fatigue from the baseline visit.
Time Frame: 4 weeks
Population: Study participants enrolled in the treatment period are included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetyl Cysteine | Placebo
Number analyzed (Participants) | 10 | 5
scores on a scale | -11.4 (14.9) | -18 (15.4)

3. Secondary Outcome: Change in Level of Blood Markers From Baseline
Description: Baseline to week 4 change in blood GSH/GSSG ratio (wherein GSH is glutathione in reduced state and GSSG is glutathione in oxidized state) and grey matter GSH concentration on 7T MR spectroscopy (MRS) between groups. We hypothesize that fatigue is associated with the GSH/GSSG ratio.
Time Frame: 4 weeks
Population: Study participants enrolled in the treatment period are included in the analysis.
Measure: Mean (Standard Deviation); unit: mean absolute change in GSH/GSSG ratio
Arm/Group | N-acetyl Cysteine | Placebo
Number analyzed (Participants) | 10 | 5
mean absolute change in GSH/GSSG ratio | -0.1 (0.6) | -0.6 (0.6)

4. Other Pre Specified Outcome: Changes in Metabolite Levels in Deep Grey Matter, and Surrounding White Matter on the Magnetic Resonance Images (MRI) From Baseline.
Description: Conventional T2/ T1-weighted images will be obtained at baseline for all subjects enrolled in the treatment phase of the study. We will perform brain MRI on 7T machine, and the sequences will be collected at baseline, and week-4 visit.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: Adverse events are collected over 4 weeks
Arm/Group | N-acetyl Cysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 6/10 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetyl Cysteine (N=10) | Placebo (N=5)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory-Other, Common cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Injury-Other, injury to back (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury-Other, Injury to face secondary to a fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT02804594/Prot_SAP_000.pdf